CLINICAL TRIAL: NCT05835258
Title: Interventional Study for the Comparison of the Oral Bioavailability of Two Melatonin Supplements
Brief Title: Oral Bioavailability of Two Melatonin Supplements
Acronym: MELFENIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: URIACH, S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MELFENIL
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Bioavailability
Keywords: Melatonin; Phenyl capsaicin; Bioenhancer
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Crossover, Randomized, Triple-Blind Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin with phenyl capsaicin (Experimental): Participants will consume one capsule of 1 mg of melatonin with phenyl capsaicin
  Interventions: Dietary Supplement: Melatonin with phenyl capsaicin
- Melatonin without phenyl capsaicin (Active Comparator): Participants will consume one capsule of 1 mg of melatonin without phenyl capsaicin
  Interventions: Dietary Supplement: Melatonin without phenyl capsaicin

INTERVENTIONS:
Dietary Supplement: Melatonin with phenyl capsaicin — Blood samples will be collected at different time points following the oral administration of the melatonin supplement with phenyl capsaicin
  Arms: Melatonin with phenyl capsaicin
Dietary Supplement: Melatonin without phenyl capsaicin — Blood samples will be collected at different time points following the oral administration of the melatonin supplement without phenyl capsaicin
  Arms: Melatonin without phenyl capsaicin

SUMMARY:
Results from several clinical studies show that orally administered melatonin has low bioavailability and a very short half-life. Phenyl capsaicin, a synthetic analogue of capsaicin, might increase its bioavailability by inhibiting the enzymes involved in its hepatic metabolism.

Thus, the hypothesis of the present study is that the administration of melatonin supplement with phenyl capsaicin presents greater bioavailability than a melatonin supplement that does not contain phenyl capsaicin.

DETAILED DESCRIPTION:
Melatonin is an endogenous indolamine that regulates many physiological functions such as reproduction, temperature, mood, bone growth or the immune system. However, since its production is closely related to the light/dark cycle, melatonin is considered one of the main chronobiotic agents that modulates circadian rhythms.

For this reason, in recent years there has been increased interest in the exogenous use of melatonin to address problems of insomnia and circadian rhythm disorders such as jet lag syndrome or shift work. Although many studies have demonstrated the effectiveness of melatonin in treating sleep disorders, pharmacokinetic studies show that it has poor oral bioavailability and a very short half-life. So, new strategies and studies are necessary to increase the low bioavailability of melatonin.

In this context, it has been shown that phenyl capsaicin, a synthetic analogue of capsaicin, might increase melatonin's bioavailability by inhibiting Cytochrome P450 liver enzymes, which are involved in its metabolism. Therefore, the main objective of this study is to quantify and compare the oral bioavailability between a melatonin supplement with phenyl capsaicin and another melatonin supplement that does not contain phenyl capsaicin.

The secondary objectives of the study are to determine the pharmacokinetic parameters:

* Maximum plasma concentration (Cmax).
* Time for maximum plasma concentration (Tmax).
* Half-life (T1/2).
* Area Under the Curve (AUC 0-inf) of plasma melatonin levels

During the study there will be 3 visits: a preselection visit (V0), a visit for the first postprandial study (V1) and after one week washing period, a visit for the second postprandial study (V2).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 65 years old.
* Sign the informed consent form.
* Know how to read, write and speak Catalan or Spanish.

Exclusion Criteria:

* Take supplements or multivitamin supplements or phytotherapeutic products that interfere with the treatment under study up to 30 days before the start of the study (e.g. L-Tryptophan or melatonin)
* Present intolerances and/or food allergies related to melatonin, phenyl capsaicin, microcrystalline cellulose or silicon dioxide .
* Be a smoker.
* Having received antibiotic treatment up to 30 days before the start of the study.
* Present values of body mass index ≤ 18kg/m^2 or ≥ 35 kg/m^2.
* Present some chronic disease with clinical manifestations: coronary heart disease, cardiovascular disease, diabetes mellitus, hypertension, ulcerative colitis, celiac disease, Crohn's disease, chronic kidney disease, cancer, benign prostatic hyperplasia, autoimmune diseases (such as fibromyalgia), respiratory and/or gastrointestinal diseases that may compromise the absorption of the compound.
* Clinical history of anemia.
* Being pregnant or intending to became pregnant.
* Be in breastfeeding period.
* Being unable to follow the study guidelines.
* Participate in or have participated in a clinical trial or nutritional intervention study in the last 30 days before inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Bioavailability of melatonin calculated by the Area Under The Curve (AUC 0-6) of plasma melatonin levels | At week 1
  Fasting melatonin levels in plasma will be determined before consuming the melatonin supplement until 6 hours postprandially at 7 points after consuming the capsule (15 min., 30 min., 45 min., 1h., 2h., 4h and 6h).
  The melatonin levels in plasma will be quantified by Liquid Chromatography coupled with Tandem Mass Spectrometry (LC-MS/MS)
Bioavailability of melatonin calculated by the Area Under The Curve (AUC 0-6) of plasma melatonin levels | At week 3
  Fasting melatonin levels in plasma will be determined before consuming the melatonin supplement until 6 hours postprandially at 7 points after consuming the capsule (15 min., 30 min., 45 min., 1h., 2h., 4h and 6h).
  The melatonin levels in plasma will be quantified by Liquid Chromatography coupled with Tandem Mass Spectrometry (LC-MS/MS)

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | At week 1
  Maximum plasma concentration of melatonin
Maximum plasma concentration (Cmax) | At week 3
  Maximum plasma concentration of melatonin
Time for maximum plasma concentration (Tmax) | At week 1
  Time period for the maximum plasma concentration of melatonin
Time for maximum plasma concentration (Tmax) | At week 3
  Time period for the maximum plasma concentration of melatonin
Half-life (T1/2) | At week 1
  Time taken for half the initial dose of melatonin administered to be eliminated from the body
Half-life (T1/2) | At week 3
  Time taken for half the initial dose of melatonin administered to be eliminated from the body
Area Under the Curve (AUC 0-inf) to infinite time of plasma melatonin levels | At week 1
  AUC 0-inf extrapolates the area to infinite time and measures the total melatonin exposure across time.
Area Under the Curve (AUC 0-inf) to infinite time of plasma melatonin levels | At week 3
  AUC 0-inf extrapolates the area to infinite time and measures the total melatonin exposure across time.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurecat, Reus, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org